CLINICAL TRIAL: NCT02033850
Title: The Rehabilitation of Attention in Patients With Mild Cognitive Impairment and Brain Subcortical Vascular Changes Using the Attention Process Training-II
Brief Title: Rehabilitation of Attention in Patients With MCI and Brain Subcortical Vascular Changes Using the APT-II
Acronym: RehAtt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Leonardo Pantoni, Full Professor of Neurology, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2010-2321706
Record Dates: First submitted 2013-12-24; First posted 2014-01-13 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-02

CONDITIONS: Mild Cognitive Impairment
Keywords: small vessel disease; cognition; treatment; rehabilitation; attention; fMRI; vascular dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia, Vascular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APT-II group (Experimental): Intervention: rehabilitation of attention using the Attention Process Training-II.
  Participants in the APT-II group will receive overall up to 40 hours of individual attention process training. Therapy will be administered in one two-hour session each week over a total of 20 weeks.
  Interventions: Behavioral: Attention Process Training-II
- standard care group (No Intervention): Participants in the standard care group will not receive cognitive training or rehabilitation interventions, will be instructed to have an usual lifestyle, and will be conventionally provided of medication and clinic consultations

INTERVENTIONS:
Behavioral: Attention Process Training-II — Rehabilitation of attention using the Attention Process Training-II
  Arms: APT-II group

SUMMARY:
Background: Subcortical Vascular Dementia (VaD), consequent to deep brain small vessel disease (SVD), is the most frequent form of VaD. The term vascular mild cognitive impairment (VMCI) defines a transitional state between normal ageing and VaD. Attentional deficits are a common finding in patients affected by VMCI or subcortical VaD. At present, no drug treatment is available to prevent vascular dementia in patients with VMCI or to improve cognitive performances of this large group of patients. Cognitive rehabilitation is directed to achieve functional changes by reinforcing, strengthening, or reestablishing previously learned patterns of behavior, or establishing new patterns of cognitive activity or compensatory mechanisms.

A hierarchical model of attention has been used to build the Attention Process Training-II (APT-II) programme.

The APT-II programme effectiveness have been demonstrated in traumatic brain injury and post-stroke rehabilitation, but there is an increasing interest in the study of cognitive rehabilitation in pathological processes that evolve over time, such as chronic cerebrovascular diseases (CVD).

Aims: The purpose of this study is to investigate whether the APT-II programme could be a useful tool in the rehabilitation of attention in individuals affected by VMCI with SVD, and if so, whether the improvement in performance is generalized to functionality in daily activities and quality of life.

Main Expected Results and Impact: Considering that the APT-II contains specific exercises to facilitate generalization to daily life, the skills that are learned by each patient during the rehabilitation programme should be generalized to daily activities.

Furthermore, the improvement of cognitive skills should also improve patient's overall quality of life because these learned skills are applicable to real-life situations. The main expected results are: 1) an impact of APT-II on disability, everyday cognition, quality of life, and performance on attention tests at short and long term after rehabilitation programme ending as compared with standard care; 2) a reduction of the risk of transition to dementia at 1 year follow-up as compared with control group.

DETAILED DESCRIPTION:
Study design

The present study is a 3-year prospective, single-blinded, randomized clinical trial. The enrolment will be carried out at the Stroke Unit and the VASCOG clinic of the Careggi University Hospital. Forty patients will be enrolled according to the following criteria: 1) MCI defined according to Winblad et al. criteria (19); 2) Evidence of impairment across attention neuropsychological tests; 3) Evidence on MRI of subcortical vascular lesions:

moderate to severe age-related white matter changes (WMC) according to a modified version of the Fazekas scale (20). Exclusion criteria: age<18 years. All enrolled patients will be evaluated at baseline according to the study protocol, that includes: 1) Clinical assessment; 2) Functional, quality of life and mood assessment; 3) Extensive neuropsychological assessment; 4) MRI protocol. After baseline assessment, participants will be randomly assigned to attention training or standard care. Stratified minimization randomization will be used to ensure the balance for possible prognostic factors (i.e., age, gender, MMSE total score, extension and localization of WMC) across the groups. All APT-II sessions will be administered by a clinical neuropsychologist, or an appositely trained graduate student in medicine. The student clinicians will receive a minimum of 30 hours of training with adult rehabilitation patients, and will be closely supervised by the neuropsychologist. Participants in the APT-II group will receive overall up to 40 hours of individual attention process training. Therapy will be administered in one two-hour session each week over a total of 20 weeks. Participants in the standard care group will not receive cognitive training or rehabilitation interventions, will be instructed to have an usual lifestyle, and will be conventionally provided of medication and clinic consultations. Each patient will be followed-up at 6 and 12 months after baseline assessment. During the follow-up visits clinical assessment, an extensive neuropsychological evaluation, and mood, functional, and quality of life assessments will be performed according to the baseline protocol. The MRI protocol will be repeated at 1-year follow-up.

Work Methodology

Baseline and follow-up clinical, neuropsychological, functional, and MRI data will be collected in a dedicated database. Data will be checked and controlled for consistency in real time during collection. At the end of the enrolment, a first exploratory data analysis will be carried out. Postprocessing of neuroimaging acquired at baseline will be performed by an experienced radiologist. At the end of each follow-up (6 and 12 months after enrollment), analysis of data (uni- and multivariate models and effect size measures) will be carried out. All analyses will be performed using SPSS 18 and will be mainly directed to: 1) evaluate the short and long-term effectiveness of the rehabilitation program, using cognitive performance and functional and quality of life measures as dependents variables (within and between groups analyses); 2) identify potential predictors of effectiveness of the rehabilitation program (multivariate model). The variables included in the model will be: demographic and vascular risk factors, baseline cognitive profile and functional status, and preexisting brain structural changes; 3) evaluate the potential protective effect of the rehabilitation program on the increase of cognitive impairment or transition to dementia at 1 year follow-up; 4) evaluate the long-term effect of rehabilitation on brain activation, using f-MRI data, whole-brain histograms, and voxel-based analyses as dependents variables (within and between groups analyses).

Milestones

* Phase 1 (4 months): 1) Project protocol establishment; 2) Dedicated database for data collection construction; 3) MRI protocol determination; 4) Training on cognitive rehabilitation
* Phase 2 (24 months): 1) Baseline patients cohort enrolment and clinical, neuropsychological, functional, and MRI data collection; 2) Neuropsychological rehabilitation program administration; 3) Follow-up assessments (6 and 12 months after enrolment)
* Phase 3 (8 months): 1) Post-processing of neuroimaging acquired at baseline and at 1-year follow-up; 2) Data completeness and consistency control; 3) Data analysis; 4) Dissemination of results

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled according to the following criteria:

* MCI defined according to Winblad et al. criteria;
* Evidence of impairment across attention neuropsychological tests;
* Evidence on MRI of subcortical vascular lesions: moderate to severe age-related white matter changes (WMC) according to a modified version of the Fazekas scale.

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Pantoni, MD, PhD, Principal Investigator — University of Milan
Locations (1):
- Stroke Unit and Neurology, VAS-COG clinic, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvadori E, Poggesi A, Valenti R, Della Rocca E, Diciotti S, Mascalchi M, Inzitari D, Pantoni L. The rehabilitation of attention in patients with mild cognitive impairment and brain subcortical vascular changes using the Attention Process Training-II. The RehAtt Study: rationale, design and methodology. Neurol Sci. 2016 Oct;37(10):1653-62. doi: 10.1007/s10072-016-2649-z. Epub 2016 Jul 1. PMID 27371187
- [Result] Pantoni L, Poggesi A, Diciotti S, Valenti R, Orsolini S, Della Rocca E, Inzitari D, Mascalchi M, Salvadori E. Effect of Attention Training in Mild Cognitive Impairment Patients with Subcortical Vascular Changes: The RehAtt Study. J Alzheimers Dis. 2017;60(2):615-624. doi: 10.3233/JAD-170428. PMID 28869475
- [Derived] Ciulli S, Citi L, Salvadori E, Valenti R, Poggesi A, Inzitari D, Mascalchi M, Toschi N, Pantoni L, Diciotti S. Prediction of Impaired Performance in Trail Making Test in MCI Patients With Small Vessel Disease Using DTI Data. IEEE J Biomed Health Inform. 2016 Jul;20(4):1026-33. doi: 10.1109/JBHI.2016.2537808. Epub 2016 Mar 3. PMID 26960231
- [Derived] Salvadori E, Poggesi A, Valenti R, Pracucci G, Pescini F, Pasi M, Nannucci S, Marini S, Del Bene A, Ciolli L, Ginestroni A, Diciotti S, Orlandi G, Di Donato I, De Stefano N, Cosottini M, Chiti A, Federico A, Dotti MT, Bonuccelli U, Inzitari D, Pantoni L; VMCI-Tuscany Study Group. Operationalizing mild cognitive impairment criteria in small vessel disease: the VMCI-Tuscany Study. Alzheimers Dement. 2016 Apr;12(4):407-18. doi: 10.1016/j.jalz.2015.02.010. Epub 2015 Jun 13. PMID 26079418

RESULTS

PARTICIPANT FLOW:
Groups:
- APT-II Group: Intervention: rehabilitation of attention using the Attention Process Training-II.
  Participants in the APT-II group received overall up to 40 hours of individual training administered in one 2-hour session each week over a total of 20 weeks.
- Standard Care Group: Participants in the standard care group did not received cognitive training or rehabilitation interventions, were instructed to have an usual lifestyle, and conventionally provided of medication and clinic consultations
Period: Overall Study
Arm/Group | APT-II Group | Standard Care Group
Started | 23 | 23
Completed | 21 | 22
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — unrelated medical reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APT-II Group | Standard Care Group | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (6) | 75.9 (7.6) | 75.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 13 | 15 | 28
Education [Mean (Standard Deviation); unit: years] | 9 (5.3) | 7.4 (3) | 8.2 (4.3)
Hypertension [Count of Participants; unit: Participants] | 18 | 20 | 38
Hypercholesterolemia [Count of Participants; unit: Participants] | 16 | 15 | 31
Diabetes [Count of Participants; unit: Participants] | 3 | 4 | 7
Smoking habits [Count of Participants; unit: Participants] — Anamnestic data: current and former smokers were included among smokers.
  Participants | 11 | 7 | 18
History of stroke [Count of Participants; unit: Participants] | 7 | 10 | 17
Alcohol consumption [Count of Participants; unit: Participants] — Current alcohol consumption considering the following three beverages: beer, wine, and liquor.
  Participants | 9 | 10 | 19
Mini Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — Total score ranging from 0 to 30: higher scores represent better performance.
  units on a scale | 27.1 (2.6) | 25.7 (3.2) | 26.4 (3)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Total score ranging from 0 to 30: higher scores represent better performance.
  units on a scale | 19.9 (4.8) | 18.6 (4.4) | 19.2 (4.6)
Activities of Daily Living (preserved items) [Mean (Standard Deviation); unit: units on a scale] — Preserved items were summed into a global score ranging from 0 (completely dependent) to 6 (completely autonomous).
  units on a scale | 5.9 (0.3) | 5.9 (0.4) | 5.9 (0.4)
Instrumental Activities of Daily Living (impaired items) [Mean (Standard Deviation); unit: units on a scale] — Impaired items were summed into a global score ranging from 0 (completely autonomous) to 8 (completely dependent).
  units on a scale | 1.9 (2.1) | 2.2 (2.4) | 2.1 (2.2)
Disability Assessment in Dementia [Mean (Standard Deviation); unit: units on a scale] — Forty dichotomous items summed into a total score and converted into a percentage ranging from 0 to 100 (higher scores represent less disability).
  units on a scale | 91.9 (11.9) | 84.2 (17.8) | 88 (15.5)
Attention Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Total score ranging from 0 (absence of attention problems) to 36 (highest presence of attention problems)
  units on a scale | 15.1 (11.5) | 15.9 (8.5) | 15.5 (9.9)
EuroQol (summary index) [Mean (Standard Deviation); unit: units on a scale] — Single summary index ranging from 0 to 1 (higher scores represent better health status)
  units on a scale | 0.7 (0.3) | 0.7 (0.3) | 0.7 (0.3)
EuroQol (visual scale) [Mean (Standard Deviation); unit: units on a scale] — Visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state)
  units on a scale | 63.1 (18.3) | 67.3 (17.5) | 65.2 (17.8)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Total score ranging from 0 (absence of depressive symptoms) to 15 (severe depressive symptoms)
  units on a scale | 4.6 (4) | 4.9 (3.8) | 4.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Functionality in Activities of Daily Living (Changes in Scores Approach)
Description: Changes in scores (Δ) approach. Delta scores (Δs) were calculated by computing the difference between the scores obtained in 2 evaluations (baseline vs. 6 months; 6 vs. 12 months; baseline vs. 12 months) for each patient. All Δs were calculated in order that a positive score indicates an improvement, while a negative score indicates a worsening. Δs were analyzed using independent sample t tests with treatment as the only independent variable.
  Scales:
  * Activities of Daily Living (ADL): preserved items summed into a global score (minimum and maximum values 0-6: higher scores mean a better outcome).
  * Instrumental Activities of Daily Living (IADL): impaired items summed into a global score (minimum and maximum values 0-8: higher scores mean a worse outcome).
  * Disability Assessment in Dementia (DAD): 40 dichotomous items summed into a total score and converted into a percentage (minimum and maximum values 0-100: higher scores mean a worse outcome).
Time Frame: Baseline, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
units on a scale
  Δs on ADL (baseline vs 6 months) | 0.1 (0.3) | 0 (0)
  Δs on ADL (6 vs 12 months) | -0.1 (0.4) | -0.2 (0.7)
  Δs on ADL (baseline vs 12 months) | 0 (0.9) | -0.2 (0.7)
  Δs on IADL (baseline vs 6 months) | -0.4 (1.1) | 0 (0.9)
  Δs on IADL (6 vs 12 months) | -0.3 (1.3) | -1 (1.7)
  Δs on IADL (baseline vs 12 months) | -0.7 (1.1) | -1 (1.7)
  Δs on DAD (baseline vs 6 months) | -2.2 (10.3) | -3.9 (11.3)
  Δs on DAD (6 vs 12 months) | -6.2 (20.2) | -3 (11.1)
  Δs on DAD (baseline vs 12 months) | -8.4 (21.1) | -6.9 (17.2)
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Δs on ADL (baseline vs 6 months); Test type: Superiority; p = .145, t-test, 2 sided
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Δs on ADL (6 vs 12 months); Test type: Superiority; p = .618, t-test, 2 sided
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Δs on ADL (baseline vs 12 months); Test type: Superiority; p = .262, t-test, 2 sided
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; Δs on IADL (baseline vs 6 months); Test type: Superiority; p = .240, t-test, 2 sided
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; Δs on IADL (6 vs 12 months); Test type: Superiority; p = .134, t-test, 2 sided
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; Δs on IADL (baseline vs 12 months); Test type: Superiority; p = .457, t-test, 2 sided
Statistical Analysis 7: Comparison: APT-II Group vs Standard Care Group; Δs on DAD (baseline vs 6 months); Test type: Superiority; p = .612, t-test, 2 sided
Statistical Analysis 8: Comparison: APT-II Group vs Standard Care Group; Δs on DAD (6 vs 12 months); Test type: Superiority; p = .522, t-test, 2 sided
Statistical Analysis 9: Comparison: APT-II Group vs Standard Care Group; Δs on DAD (baseline vs 12 months); Test type: Superiority; p = .800, t-test, 2 sided

2. Primary Outcome: Quality of Life (Changes in Scores Approach)
Description: Changes in scores (Δ) approach. Delta scores (Δs) were calculated by computing the difference between the scores obtained in 2 evaluations (baseline vs. 6 months; 6 vs. 12 months; baseline vs. 12 months) for each patient. All Δs were calculated in order that a positive score indicates an improvement, while a negative score indicates a worsening. Δs were analyzed using independent sample t tests with treatment as the only independent variable.
  Scales:
  * Short Form Health Survey summary scores: Physical and Mental Component Summary (PCS, MCS) (minimum and maximum values 0-100: lower scores mean worse outcome).
  * EuroQol (EQ): summary index (min-max values 0-1) and visual analogue scale (minimum and maximum values 0-100: higher scores mean better outcome).
  * Attention Questionnaire (AQ) total score (minimum and maximum values 0-36: higher scores mean worse outcome).
  * Geriatric Depression Scale (GDS) total score (minimum and maximum values 0-15: higher scores mean worse outcome).
Time Frame: Baseline, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
units on a scale
  Δs on AQ (baseline vs 6 months) | -1.3 (7.8) | 2.1 (9.3)
  Δs on AQ (6 vs 12 months) | -3.8 (7.9) | -3.3 (5)
  Δs on AQ (baseline vs 12 months) | -5.1 (8.4) | -1.2 (10.6)
  Δs on EQ index (baseline vs 6 months) | 0.1 (0.2) | 0.1 (0.2)
  Δs on EQ index (6 vs 12 months) | -0.1 (0.2) | 0 (0.2)
  Δs on EQ index (baseline vs 12 months) | 0 (0.3) | 0.1 (0.3)
  Δs on EQ visual (baseline vs 6 months) | 5.2 (15.3) | -2.3 (9.2)
  Δs on EQ visual (6 vs 12 months) | -0.2 (12.9) | -2 (15.8)
  Δs on EQ visual (baseline vs 12 months) | 5 (14.2) | -4.3 (16.6)
  Δs on GDS (baseline vs 6 months) | -0.1 (2.1) | -0.8 (2.9)
  Δs on GDS (6 vs 12 months) | 0 (2.7) | 0 (2.9)
  Δs on GDS (baseline vs 12 months) | -0.1 (2.9) | -0.7 (2.5)
  Δs on MCS (baseline vs 6 months) | 1.4 (5.3) | 3 (11.4)
  Δs on MCS (6 vs 12 months) | -0.1 (6.2) | -2.8 (9.3)
  Δs on MCS (baseline vs 12 months) | 1.3 (7) | 0.2 (9.6)
  Δs on PCS (baseline vs 6 months) | -1.1 (6.5) | -1.9 (8.2)
  Δs on PCS (6 vs 12 months) | -0.9 (6.6) | 0.5 (8.3)
  Δs on PCS (baseline vs 12 months) | -2 (8.1) | -1.5 (10.2)
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Δs on AQ (baseline vs 6 months); Test type: Superiority; p = .204, t-test, 2 sided
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Δs on AQ (6 vs 12 months); Test type: Superiority; p = .810, t-test, 2 sided
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Δs on AQ (baseline vs 12 months); Test type: Superiority; p = .193, t-test, 2 sided
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; Δs on EQ index (baseline vs 6 months); Test type: Superiority; p = .698, t-test, 2 sided
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; Δs on EQ index (6 vs 12 months); Test type: Superiority; p = .283, t-test, 2 sided
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; Δs on EQ index (baseline vs 12 months); Test type: Superiority; p = .647, t-test, 2 sided
Statistical Analysis 7: Comparison: APT-II Group vs Standard Care Group; Δs on EQ visual (baseline vs 6 months); Test type: Superiority; p = .057, t-test, 2 sided
Statistical Analysis 8: Comparison: APT-II Group vs Standard Care Group; Δs on EQ visual (6 vs 12 months); Test type: Superiority; p = .685, t-test, 2 sided
Statistical Analysis 9: Comparison: APT-II Group vs Standard Care Group; Δs on EQ visual (baseline vs 12 months); Test type: Superiority; p = .056, t-test, 2 sided
Statistical Analysis 10: Comparison: APT-II Group vs Standard Care Group; Δs on GDS (baseline vs 6 months); Test type: Superiority; p = .393, t-test, 2 sided
Statistical Analysis 11: Comparison: APT-II Group vs Standard Care Group; Δs on GDS (6 vs 12 months); Test type: Superiority; p = .958, t-test, 2 sided
Statistical Analysis 12: Comparison: APT-II Group vs Standard Care Group; Δs on GDS (baseline vs 12 months); Test type: Superiority; p = .448, t-test, 2 sided
Statistical Analysis 13: Comparison: APT-II Group vs Standard Care Group; Δs on MCS (baseline vs 6 months); Test type: Superiority; p = .567, t-test, 2 sided
Statistical Analysis 14: Comparison: APT-II Group vs Standard Care Group; Δs on MCS (6 vs 12 months); Test type: Superiority; p = .274, t-test, 2 sided
Statistical Analysis 15: Comparison: APT-II Group vs Standard Care Group; Δs on MCS (baseline vs 12 months); Test type: Superiority; p = .668, t-test, 2 sided
Statistical Analysis 16: Comparison: APT-II Group vs Standard Care Group; Δs on PCS (baseline vs 6 months); Test type: Superiority; p = .709, t-test, 2 sided
Statistical Analysis 17: Comparison: APT-II Group vs Standard Care Group; Δs on PCS (6 vs 12 months); Test type: Superiority; p = .567, t-test, 2 sided
Statistical Analysis 18: Comparison: APT-II Group vs Standard Care Group; Δs on PCS (baseline vs 12 months); Test type: Superiority; p = .867, t-test, 2 sided

3. Primary Outcome: Quality of Life (Clinically Significance Approach)
Description: Clinically significance approach. The availability of t scores for the Short Form Health Survey (SF-36) Physical and Mental Component Summary scores (MCS, PCS) allowed us to classify each patient evaluation as 'normal well-being' (t score >40) or 'reduced well-being' (t score ≤40) at each visit (higher scores mean a better outcome). Variations in performance categories over time (baseline vs. 6 month; 6 vs. 12 month; baseline vs. 12 month) were evaluated for each patient and dichotomized as: 'stable or better evaluation' or 'worst evaluation'. Variations in performance categories were analyzed using chi square tests.
Time Frame: Baseline, 6 months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
Participants
  MCS outcome (baseline vs 6 months): Stable/better | 19 | 19
  MCS outcome (baseline vs 6 months): Worse | 2 | 3
  MCS outcome (6 vs 12 months): Stable/better | 18 | 18
  MCS outcome (6 vs 12 months): Worse | 3 | 4
  MCS outcome (baseline vs 12 months): Stable/better | 18 | 17
  MCS outcome (baseline vs 12 months): Worse | 3 | 5
  PCS outcome (baseline vs 6 months): Stable/better | 16 | 17
  PCS outcome (baseline vs 6 months): Worse | 5 | 5
  PCS outcome (6 vs 12 months): Stable/better | 16 | 20
  PCS outcome (6 vs 12 months): Worse | 5 | 2
  PCS outcome (baseline vs 12 months): Stable/better | 14 | 17
  PCS outcome (baseline vs 12 months): Worse | 7 | 5
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; MCS outcome (baseline vs 6 months); Test type: Superiority; p = .095, Chi-squared
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; MCS outcome (6 vs 12 months); Test type: Superiority; p = .729, Chi-squared
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; MCS outcome (baseline vs 12 months); Test type: Superiority; p = .115, Chi-squared
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; PCS outcome (baseline vs 6 months); Test type: Superiority; p = .576, Chi-squared
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; PCS outcome (6 vs 12 months); Test type: Superiority; p = .191, Chi-squared
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; PCS outcome (baseline vs 12 months); Test type: Superiority; p = .790, Chi-squared

4. Secondary Outcome: Cognitive Performance (Changes in Scores Approach)
Description: Delta (Δ) scores were calculated by computing the difference between the scores obtained in 2 evaluations (baseline vs. 6 months; 6 vs. 12 months; baseline vs. 12 months) for each patient. A positive Δ score indicates an improvement, while a negative Δ score indicates a worsening. Delta scores were analyzed using independent sample t tests with treatment as the only independent variable.
  Test battery: Montreal Cognitive Assessment MoCA (minimum and maximum values 0-30); Mini Mental Status Examination MMSE (minimum and maximum values 0-30), Rey Auditory-Verbal Learning RAVL immediate (minimum and maximum values 0-75) and recall (minimum and maximum values 0-15), Short story (minimum and maximum values 0-28), Rey-Osterrieth Complex Figure ROCF copy and recall (minimum and maximum values 0-36), Visual search (minimum and maximum values 0-50), Symbol Digit Modalities Test SDMT (minimum and maximum values 0-110). Higher scores mean better outcome for all tests.
Time Frame: Baseline, 6 months and 12 months
Population: Not all the participants completed the entire neuropsychological evaluation during the follow-up visits due to refuse or failure to learn or remember the instructions, or to perform the task until the end
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
units on a scale
  Δs on MoCA (baseline vs 6 months): number analyzed (Participants) | 20 | 22
  Δs on MoCA (baseline vs 6 months) | 1.1 (4.1) | 1.1 (3.4)
  Δs on MoCA (6 vs 12 months) | 0.8 (3) | -0.3 (2.7)
  Δs on MoCA (baseline vs 12 months): number analyzed (Participants) | 20 | 22
  Δs on MoCA (baseline vs 12 months) | 2 (3.9) | 0.8 (4.5)
  Δs on MMSE (baseline vs 6 months) | -0.3 (1.9) | -0.8 (1.9)
  Δs on MMSE (6 vs 12 months) | -0.4 (2.6) | 0.4 (1.9)
  Δs on MMSE (baseline vs 12 months) | -0.7 (2.8) | -0.3 (1.8)
  Δs on RAVL immediate (baseline vs 6 months) | 2 (7.6) | 1.6 (4.9)
  Δs on RAVL immediate (6 vs 12 months) | 1.8 (4.9) | -1.4 (3.8)
  Δs on RAVL immediate (baseline vs 12 months) | 3.8 (6.1) | 0.2 (4.4)
  Δs on RAVL recall (baseline vs 6 months) | 0.3 (2.2) | 0.4 (2.5)
  Δs on RAVL recall (6 vs 12 months) | 0.5 (2.5) | -0.3 (2)
  Δs on RAVL recall (baseline vs 12 months) | 0.9 (2.3) | 0.1 (2)
  Δs on ROCF recall (baseline vs 6 months): number analyzed (Participants) | 18 | 21
  Δs on ROCF recall (baseline vs 6 months) | -0.4 (7.4) | 2.3 (6.7)
  Δs on ROCF recall (6 vs 12 months): number analyzed (Participants) | 16 | 20
  Δs on ROCF recall (6 vs 12 months) | 0.6 (6.5) | -1 (3.7)
  Δs on ROCF recall (baseline vs 12 months): number analyzed (Participants) | 17 | 20
  Δs on ROCF recall (baseline vs 12 months) | 0.7 (9.7) | 1.5 (5.8)
  Δs on short story (baseline vs 6 months) | -1.3 (3.1) | -0.1 (2.5)
  Δs on short story (6 vs 12 months) | 0.7 (2.2) | 0 (2.9)
  Δs on short story (baseline vs 12 months) | -0.7 (2.7) | -0.1 (3.2)
  Δs on visual search (baseline vs 6 months): number analyzed (Participants) | 21 | 21
  Δs on visual search (baseline vs 6 months) | -3.4 (7.1) | -2.6 (9.1)
  Δs on visual search (6 vs 12 months): number analyzed (Participants) | 21 | 21
  Δs on visual search (6 vs 12 months) | 0.3 (6.9) | -1.5 (7.3)
  Δs on visual search (baseline vs 12 months): number analyzed (Participants) | 21 | 20
  Δs on visual search (baseline vs 12 months) | -3 (8.2) | -4.2 (9.7)
  Δs on SDMT (baseline vs 6 months) | 1.1 (5.4) | -0.3 (4.1)
  Δs on SDMT (6 vs 12 months) | -2 (6.1) | 0.3 (5.8)
  Δs on SDMT (baseline vs 12 months) | -0.9 (4.6) | -0.1 (7.8)
  Δs on ROCF copy (baseline vs 6 months): number analyzed (Participants) | 20 | 22
  Δs on ROCF copy (baseline vs 6 months) | -1.5 (7.9) | 2.3 (6.7)
  Δs on ROCF copy (6 vs 12 months): number analyzed (Participants) | 19 | 21
  Δs on ROCF copy (6 vs 12 months) | -0.3 (6.1) | -2.8 (7.3)
  Δs on ROCF copy (baseline vs 12 months): number analyzed (Participants) | 20 | 21
  Δs on ROCF copy (baseline vs 12 months) | -1.6 (8.8) | -0.9 (7.8)
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Δs on MoCA (baseline vs 6 months); Test type: Superiority; p = .936, t-test, 2 sided
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Δs on MoCA (6 vs 12 months); Test type: Superiority; p = .188, t-test, 2 sided
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Δs on MoCA (baseline vs 12 months); Test type: Superiority; p = .381, t-test, 2 sided
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; Δs on MMSE (baseline vs 6 months); Test type: Superiority; p = .458, t-test, 2 sided
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; Δs on MMSE (6 vs 12 months); Test type: Superiority; p = .236, t-test, 2 sided
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; Δs on MMSE (baseline vs 12 months); Test type: Superiority; p = .601, t-test, 2 sided
Statistical Analysis 7: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL immediate (baseline vs 6 months); Test type: Superiority; p = .839, t-test, 2 sided
Statistical Analysis 8: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL immediate (6 vs 12 months); Test type: Superiority; p = .021, t-test, 2 sided
Statistical Analysis 9: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL immediate (baseline vs 12 months); Test type: Superiority; p = .032, t-test, 2 sided
Statistical Analysis 10: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL recall (baseline vs 6 months); Test type: Superiority; p = .858, t-test, 2 sided
Statistical Analysis 11: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL recall (6 vs 12 months); Test type: Superiority; p = .212, t-test, 2 sided
Statistical Analysis 12: Comparison: APT-II Group vs Standard Care Group; Δs on RAVL recall (baseline vs 12 months); Test type: Superiority; p = .268, t-test, 2 sided
Statistical Analysis 13: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF recall (baseline vs 6 months); Test type: Superiority; p = .184, t-test, 2 sided
Statistical Analysis 14: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF recall (6 vs 12 months); Test type: Superiority; p = .358, t-test, 2 sided
Statistical Analysis 15: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF recall (baseline vs 12 months); Test type: Superiority; p = .768, t-test, 2 sided
Statistical Analysis 16: Comparison: APT-II Group vs Standard Care Group; Δs on short story (baseline vs 6 months); Test type: Superiority; p = .164, t-test, 2 sided
Statistical Analysis 17: Comparison: APT-II Group vs Standard Care Group; Δs on short story (6 vs 12 months); Test type: Superiority; p = .420, t-test, 2 sided
Statistical Analysis 18: Comparison: APT-II Group vs Standard Care Group; Δs on short story (baseline vs 12 months); Test type: Superiority; p = .527, t-test, 2 sided
Statistical Analysis 19: Comparison: APT-II Group vs Standard Care Group; Δs on visual search (baseline vs 6 months); Test type: Superiority; p = .762, t-test, 2 sided
Statistical Analysis 20: Comparison: APT-II Group vs Standard Care Group; Δs on visual search (6 vs 12 months); Test type: Superiority; p = .405, t-test, 2 sided
Statistical Analysis 21: Comparison: APT-II Group vs Standard Care Group; Δs on visual search (baseline vs 12 months); Test type: Superiority; p = .674, t-test, 2 sided
Statistical Analysis 22: Comparison: APT-II Group vs Standard Care Group; Δs on SDMT (baseline vs 6 months); Test type: Superiority; p = .328, t-test, 2 sided
Statistical Analysis 23: Comparison: APT-II Group vs Standard Care Group; Δs on SDMT (6 vs 12 months); Test type: Superiority; p = .198, t-test, 2 sided
Statistical Analysis 24: Comparison: APT-II Group vs Standard Care Group; Δs on SDMT (baseline vs 12 months); Test type: Superiority; p = .639, t-test, 2 sided
Statistical Analysis 25: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF copy (baseline vs 6 months); Test type: Superiority; p = .098, t-test, 2 sided
Statistical Analysis 26: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF copy (6 vs 12 months); Test type: Superiority; p = .235, t-test, 2 sided
Statistical Analysis 27: Comparison: APT-II Group vs Standard Care Group; Δs on ROCF copy (baseline vs 12 months); Test type: Superiority; p = .789, t-test, 2 sided

5. Secondary Outcome: Cognitive Performance TMT-A, TMT-B, Stroop (Changes in Scores Approach)
Description: Delta (Δ) scores were calculated by computing the difference between the scores obtained in 2 evaluations (baseline vs. 6 months; 6 vs. 12 months; baseline vs. 12 months) for each patient. A positive Δ score indicates an improvement, while a negative Δ score indicates a worsening. Delta scores were analyzed using independent sample t tests with treatment as the only independent variable.
  Cognitive tests based on execution time in seconds: Trail Making Test TMT part A (minimum and maximum values 0-300), TMT part B (minimum and maximum values 0-300), and Stroop Test (minimum and maximum values 0-300). Higher scores mean worse outcome.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
seconds
  Δs on Stroop test (baseline vs 6 months) | 0.4 (16.4) | -1.7 (25.2)
  Δs on Stroop test (6 vs 12 months) | 1.7 (15.3) | -3.4 (25.6)
  Δs on Stroop test (baseline vs 12 months) | 2.2 (18.4) | -5.1 (26)
  Δs on TMT-A (baseline vs 6 months) | -7.7 (23.8) | 3.9 (28.2)
  Δs on TMT-A (6 vs 12 months) | 2.9 (24.6) | -11.83 (30.7)
  Δs on TMT-A (baseline vs 12 months) | -4.8 (29.6) | -13.2 (44.9)
  Δs on TMT-B (baseline vs 6 months) | 24.5 (55.9) | -14.1 (48.5)
  Δs on TMT-B (6 vs 12 months) | -13.2 (51.4) | -4.2 (21)
  Δs on TMT-B (baseline vs 12 months) | 10.7 (45.3) | -4.6 (53.8)
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Δs on Stroop test (baseline vs 6 months); Test type: Superiority; p = .743, t-test, 2 sided
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Δs on Stroop test (6 vs 12 months); Test type: Superiority; p = .428, t-test, 2 sided
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Δs on Stroop test (baseline vs 12 months); Test type: Superiority; p = .294, t-test, 2 sided
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-A (baseline vs 6 months); Test type: Superiority; p = .157, t-test, 2 sided
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-A (6 vs 12 months); Test type: Superiority; p = .094, t-test, 2 sided
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-A (baseline vs 12 months); Test type: Superiority; p = .476, t-test, 2 sided
Statistical Analysis 7: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-B (baseline vs 6 months); Test type: Superiority; p = .142, t-test, 2 sided
Statistical Analysis 8: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-B (6 vs 12 months); Test type: Superiority; p = .651, t-test, 2 sided
Statistical Analysis 9: Comparison: APT-II Group vs Standard Care Group; Δs on TMT-B (baseline vs 12 months); Test type: Superiority; p = .534, t-test, 2 sided

6. Secondary Outcome: Cognitive Performance Verbal Fluency (Changes in Scores Approach)
Description: Delta (Δ) scores were calculated by computing the difference between the scores obtained in 2 evaluations (baseline vs. 6 months; 6 vs. 12 months; baseline vs. 12 months) for each patient. A positive Δ score indicates an improvement, while a negative Δ score indicates a worsening. Delta scores were analyzed using independent sample t tests with treatment as the only independent variable.
  Cognitive tests based on the total number of words produced: phonemic (minimum and maximum values not applicable) and semantic verbal fluency (minimum and maximum values not applicable). Higher scores mean better outcome for both tests.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: words
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
words
  Δs on phonemic fluency (baseline vs 6 months) | 0 (6.7) | 0.3 (5.4)
  Δs on phonemic fluency (6 vs 12 months) | 0.1 (6.4) | -0.3 (6.5)
  Δs on phonemic fluency (baseline vs 12 months) | 0.1 (7.7) | 0 (6.7)
  Δs on semantic fluency (baseline vs 6 months) | -0.5 (5.3) | 0.8 (5)
  Δs on semantic fluency (6 vs 12 months) | -0.1 (5.9) | 0 (5.6)
  Δs on semantic fluency (baseline vs 12 months) | -0.6 (7.2) | 0.8 (5.9)
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Δs on phonemic fluency (baseline vs 6 months); Test type: Superiority; p = .882, t-test, 2 sided
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Δs on phonemic fluency (6 vs 12 months); Test type: Superiority; p = .835, t-test, 2 sided
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Δs on phonemic fluency (baseline vs 12 months); Test type: Superiority; p = .951, t-test, 2 sided
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; Δs on semantic fluency (baseline vs 6 months); Test type: Superiority; p = .392, t-test, 2 sided
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; Δs on semantic fluency (6 vs 12 months); Test type: Superiority; p = .973, t-test, 2 sided
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; Δs on semantic fluency (baseline vs 12 months); Test type: Superiority; p = .486, t-test, 2 sided

7. Secondary Outcome: Cognitive Performance (Clinically Significance Approach)
Description: Clinically significance approach. The availability of national norms for the cognitive variables allowed us to classify each patient's performance as 'normal', 'borderline' or 'abnormal' at each visit. Variations in performance categories over time (baseline vs. 6 month; 6 vs. 12 month; baseline vs. 12 month) were evaluated for each patient and dichotomized as: 'stable or better evaluation' or 'worst evaluation'. Variations in performance categories were analyzed using chi square tests.
  Test battery:
  * global cognitive functioning: Montreal Cognitive Assessment, MoCA; Mini Mental Status Examination, MMSE
  * memory: Rey Auditory-Verbal Learning (RAVL) immediate and recall, Short story, Rey-Osterrieth Complex Figure (ROCF) recall
  * attention/executive function: Trail Making Test part A and B (TMT-A and B), Visual search, Symbol Digit Modalities Test (SDMT), Stroop Test
  * language: phonemic and semantic verbal fluency
  * constructional praxis: ROCF copy
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
Participants
  MoCA variations (baseline vs 6 months): number analyzed (Participants) | 20 | 22
  MoCA variations (baseline vs 6 months): Stable/better | 18 | 20
  MoCA variations (baseline vs 6 months): Worst | 2 | 2
  MoCA variations (6 vs 12 months): Stable/better | 20 | 18
  MoCA variations (6 vs 12 months): Worst | 1 | 4
  MoCA variations (baseline vs 12 months): number analyzed (Participants) | 20 | 22
  MoCA variations (baseline vs 12 months): Stable/better | 18 | 19
  MoCA variations (baseline vs 12 months): Worst | 2 | 3
  MMSE variations (baseline vs 6 months): Stable/better | 20 | 21
  MMSE variations (baseline vs 6 months): Worst | 1 | 1
  MMSE variations (6 vs 12 months): Stable/better | 20 | 21
  MMSE variations (6 vs 12 months): Worst | 1 | 1
  MMSE variations (baseline vs 12 months): Stable/better | 20 | 22
  MMSE variations (baseline vs 12 months): Worst | 1 | 0
  RAVL immed. variations (baseline vs 6 months): Stable/better | 16 | 21
  RAVL immed. variations (baseline vs 6 months): Worst | 5 | 1
  RAVL immed. variations (6 vs 12 months): Stable/better | 20 | 17
  RAVL immed. variations (6 vs 12 months): Worst | 1 | 5
  RAVL immed. variations (baseline vs 12 months): Stable/better | 19 | 17
  RAVL immed. variations (baseline vs 12 months): Worst | 2 | 5
  RAVL recall variations (baseline vs 6 months): Stable/better | 20 | 17
  RAVL recall variations (baseline vs 6 months): Worst | 1 | 5
  RAVL recall variations (6 vs 12 months): Stable/better | 20 | 18
  RAVL recall variations (6 vs 12 months): Worst | 1 | 4
  RAVL recall variations (baseline vs 12 months): Stable/better | 19 | 18
  RAVL recall variations (baseline vs 12 months): Worst | 2 | 4
  ROCF recall variations (baseline vs 6 months): number analyzed (Participants) | 18 | 21
  ROCF recall variations (baseline vs 6 months): Stable/better | 13 | 16
  ROCF recall variations (baseline vs 6 months): Worst | 5 | 5
  ROCF recall variations (6 vs 12 months): number analyzed (Participants) | 16 | 20
  ROCF recall variations (6 vs 12 months): Stable/better | 15 | 15
  ROCF recall variations (6 vs 12 months): Worst | 1 | 5
  ROCF recall variations (baseline vs 12 months): number analyzed (Participants) | 17 | 20
  ROCF recall variations (baseline vs 12 months): Stable/better | 15 | 16
  ROCF recall variations (baseline vs 12 months): Worst | 2 | 4
  Short story variations (baseline vs 6 months): Stable/better | 17 | 18
  Short story variations (baseline vs 6 months): Worst | 4 | 4
  Short story variations (6 vs 12 months): Stable/better | 20 | 20
  Short story variations (6 vs 12 months): Worst | 1 | 2
  Short story variations (baseline vs 12 months): Stable/better | 19 | 18
  Short story variations (baseline vs 12 months): Worst | 2 | 4
  Visual search variations (baseline vs 6 months): number analyzed (Participants) | 21 | 21
  Visual search variations (baseline vs 6 months): Stable/better | 15 | 15
  Visual search variations (baseline vs 6 months): Worst | 6 | 6
  Visual search variations (6 vs 12 months): number analyzed (Participants) | 21 | 21
  Visual search variations (6 vs 12 months): Stable/better | 20 | 15
  Visual search variations (6 vs 12 months): Worst | 1 | 6
  Visual search variations (baseline vs 12 months): number analyzed (Participants) | 21 | 20
  Visual search variations (baseline vs 12 months): Stable/better | 15 | 13
  Visual search variations (baseline vs 12 months): Worst | 6 | 7
  SDMT variations (baseline vs 6 months): Stable/better | 19 | 21
  SDMT variations (baseline vs 6 months): Worst | 2 | 1
  SDMT variations (6 vs 12 months): Stable/better | 19 | 19
  SDMT variations (6 vs 12 months): Worst | 2 | 3
  SDMT variations (baseline vs 12 months): Stable/better | 20 | 18
  SDMT variations (baseline vs 12 months): Worst | 1 | 4
  Stroop test variations (baseline vs 6 months): Stable/better | 19 | 20
  Stroop test variations (baseline vs 6 months): Worst | 2 | 2
  Stroop test variations (6 vs 12 months): Stable/better | 19 | 18
  Stroop test variations (6 vs 12 months): Worst | 2 | 4
  Stroop test variations (baseline vs 12 months): Stable/better | 18 | 17
  Stroop test variations (baseline vs 12 months): Worst | 3 | 5
  TMT-A variations (baseline vs 6 months): Stable/better | 15 | 18
  TMT-A variations (baseline vs 6 months): Worst | 6 | 4
  TMT-A variations (6 vs 12 months): Stable/better | 19 | 17
  TMT-A variations (6 vs 12 months): Worst | 2 | 5
  TMT-A variations (baseline vs 12 months): Stable/better | 18 | 16
  TMT-A variations (baseline vs 12 months): Worst | 3 | 6
  TMT-B variations (baseline vs 6 months): number analyzed (Participants) | 18 | 20
  TMT-B variations (baseline vs 6 months): Stable/better | 16 | 16
  TMT-B variations (baseline vs 6 months): Worst | 2 | 4
  TMT-B variations (6 vs 12 months): number analyzed (Participants) | 18 | 17
  TMT-B variations (6 vs 12 months): Stable/better | 16 | 15
  TMT-B variations (6 vs 12 months): Worst | 2 | 2
  TMT-B variations (baseline vs 12 months): number analyzed (Participants) | 19 | 17
  TMT-B variations (baseline vs 12 months): Stable/better | 16 | 14
  TMT-B variations (baseline vs 12 months): Worst | 3 | 3
  Phonemic fluency variations (baseline vs 6 months): Stable/better | 19 | 18
  Phonemic fluency variations (baseline vs 6 months): Worst | 2 | 4
  Phonemic fluency variations (6 vs 12 months): Stable/better | 19 | 20
  Phonemic fluency variations (6 vs 12 months): Worst | 2 | 2
  Phonemic fluency variation (baseline vs 12 months): Stable/better | 18 | 19
  Phonemic fluency variation (baseline vs 12 months): Worst | 3 | 3
  Semantic fluency variations (baseline vs 6 months): Stable/better | 18 | 19
  Semantic fluency variations (baseline vs 6 months): Worst | 3 | 3
  Semantic fluency variations (6 vs 12 months): Stable/better | 19 | 19
  Semantic fluency variations (6 vs 12 months): Worst | 2 | 3
  Semantic fluency variation (baseline vs 12 months): Stable/better | 18 | 19
  Semantic fluency variation (baseline vs 12 months): Worst | 3 | 3
  ROCF copy variations (baseline vs 6 months): number analyzed (Participants) | 20 | 22
  ROCF copy variations (baseline vs 6 months): Stable/better | 20 | 22
  ROCF copy variations (baseline vs 6 months): Worst | 0 | 0
  ROCF copy variations (6 vs 12 months): number analyzed (Participants) | 19 | 21
  ROCF copy variations (6 vs 12 months): Stable/better | 18 | 14
  ROCF copy variations (6 vs 12 months): Worst | 1 | 7
  ROCF copy variations (baseline vs 12 months): number analyzed (Participants) | 20 | 21
  ROCF copy variations (baseline vs 12 months): Stable/better | 19 | 17
  ROCF copy variations (baseline vs 12 months): Worst | 1 | 4
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; MoCA variations (baseline vs 6 months); Test type: Superiority; p = .920, Chi-squared
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; MoCA variations (6 vs 12 months); Test type: Superiority; p = .170, Chi-squared
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; MoCA variations (baseline vs 12 months); Test type: Superiority; p = .716, Chi-squared
Statistical Analysis 4: Comparison: APT-II Group vs Standard Care Group; MMSE variations (baseline vs 6 months); Test type: Superiority; p = .973, Chi-squared
Statistical Analysis 5: Comparison: APT-II Group vs Standard Care Group; MMSE variations (6 vs 12 months); Test type: Superiority; p = .973, Chi-squared
Statistical Analysis 6: Comparison: APT-II Group vs Standard Care Group; MMSE variations (baseline vs 12 months); Test type: Superiority; p = .300, Chi-squared
Statistical Analysis 7: Comparison: APT-II Group vs Standard Care Group; RAVL immed. variations (baseline vs 6 months); Test type: Superiority; p = .068, Chi-squared
Statistical Analysis 8: Comparison: APT-II Group vs Standard Care Group; RAVL immed. variations (6 vs 12 months); Test type: Superiority; p = .089, Chi-squared
Statistical Analysis 9: Comparison: APT-II Group vs Standard Care Group; RAVL immed. variations (baseline vs 12 months); Test type: Superiority; p = .241, Chi-squared
Statistical Analysis 10: Comparison: APT-II Group vs Standard Care Group; RAVL recall variations (baseline vs 6 months); Test type: Superiority; p = .089, Chi-squared
Statistical Analysis 11: Comparison: APT-II Group vs Standard Care Group; RAVL recall variations (6 vs 12 months); Test type: Superiority; p = .170, Chi-squared
Statistical Analysis 12: Comparison: APT-II Group vs Standard Care Group; RAVL recall variations (baseline vs 12 months); Test type: Superiority; p = .413, Chi-squared
Statistical Analysis 13: Comparison: APT-II Group vs Standard Care Group; ROCF recall variations (baseline vs 6 months); Test type: Superiority; p = .777, Chi-squared
Statistical Analysis 14: Comparison: APT-II Group vs Standard Care Group; ROCF recall variations (6 vs 12 months); Test type: Superiority; p = .134, Chi-squared
Statistical Analysis 15: Comparison: APT-II Group vs Standard Care Group; ROCF recall variations (baseline vs 12 months); Test type: Superiority; p = .498, Chi-squared
Statistical Analysis 16: Comparison: APT-II Group vs Standard Care Group; Short story variations (baseline vs 6 months); Test type: Superiority; p = .942, Chi-squared
Statistical Analysis 17: Comparison: APT-II Group vs Standard Care Group; Short story variations (6 vs 12 months); Test type: Superiority; p = .578, Chi-squared
Statistical Analysis 18: Comparison: APT-II Group vs Standard Care Group; Short story variations (baseline vs 12 months); Test type: Superiority; p = .413, Chi-squared
Statistical Analysis 19: Comparison: APT-II Group vs Standard Care Group; Visual search variations (baseline vs 6 months); Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 20: Comparison: APT-II Group vs Standard Care Group; Visual search variations (6 vs 12 months); Test type: Superiority; p = .038, Chi-squared
Statistical Analysis 21: Comparison: APT-II Group vs Standard Care Group; Visual search variations (baseline vs 12 months); Test type: Superiority; p = .658, Chi-squared
Statistical Analysis 22: Comparison: APT-II Group vs Standard Care Group; SDMT variations (baseline vs 6 months); Test type: Superiority; p = .522, Chi-squared
Statistical Analysis 23: Comparison: APT-II Group vs Standard Care Group; SDMT variations (6 vs 12 months); Test type: Superiority; p = .674, Chi-squared
Statistical Analysis 24: Comparison: APT-II Group vs Standard Care Group; SDMT variations (baseline vs 12 months); Test type: Superiority; p = .170, Chi-squared
Statistical Analysis 25: Comparison: APT-II Group vs Standard Care Group; Stroop test variations (baseline vs 6 months); Test type: Superiority; p = .961, Chi-squared
Statistical Analysis 26: Comparison: APT-II Group vs Standard Care Group; Stroop test variations (6 vs 12 months); Test type: Superiority; p = .413, Chi-squared
Statistical Analysis 27: Comparison: APT-II Group vs Standard Care Group; Stroop test variations (baseline vs 12 months); Test type: Superiority; p = .477, Chi-squared
Statistical Analysis 28: Comparison: APT-II Group vs Standard Care Group; TMT-A variations (baseline vs 6 months); Test type: Superiority; p = .420, Chi-squared
Statistical Analysis 29: Comparison: APT-II Group vs Standard Care Group; TMT-A variations (6 vs 12 months); Test type: Superiority; p = .241, Chi-squared
Statistical Analysis 30: Comparison: APT-II Group vs Standard Care Group; TMT-A variations (baseline vs 12 months); Test type: Superiority; p = .295, Chi-squared
Statistical Analysis 31: Comparison: APT-II Group vs Standard Care Group; TMT-B variations (baseline vs 6 months); Test type: Superiority; p = .453, Chi-squared
Statistical Analysis 32: Comparison: APT-II Group vs Standard Care Group; TMT-B variations (6 vs 12 months); Test type: Superiority; p = .952, Chi-squared
Statistical Analysis 33: Comparison: APT-II Group vs Standard Care Group; TMT-B variations (baseline vs 12 months); Test type: Superiority; p = .881, Chi-squared
Statistical Analysis 34: Comparison: APT-II Group vs Standard Care Group; Phonemic fluency variations (baseline vs 6 months); Test type: Superiority; p = .413, Chi-squared
Statistical Analysis 35: Comparison: APT-II Group vs Standard Care Group; Phonemic fluency variations (6 vs 12 months); Test type: Superiority; p = .961, Chi-squared
Statistical Analysis 36: Comparison: APT-II Group vs Standard Care Group; Phonemic fluency variation (baseline vs 12 months); Test type: Superiority; p = .951, Chi-squared
Statistical Analysis 37: Comparison: APT-II Group vs Standard Care Group; Semantic fluency variations (baseline vs 6 months); Test type: Superiority; p = .951, Chi-squared
Statistical Analysis 38: Comparison: APT-II Group vs Standard Care Group; Semantic fluency variations (6 vs 12 months); Test type: Superiority; p = .674, Chi-squared
Statistical Analysis 39: Comparison: APT-II Group vs Standard Care Group; Semantic fluency variation (baseline vs 12 months); Test type: Superiority; p = .951, Chi-squared
Statistical Analysis 40: Comparison: APT-II Group vs Standard Care Group; ROCF copy variations (baseline vs 6 months); Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 41: Comparison: APT-II Group vs Standard Care Group; ROCF copy variations (6 vs 12 months); Test type: Superiority; p = .027, Chi-squared
Statistical Analysis 42: Comparison: APT-II Group vs Standard Care Group; ROCF copy variations (baseline vs 12 months); Test type: Superiority; p = .169, Chi-squared

8. Secondary Outcome: Transition to Dementia
Description: Data collected during the 1-year follow-up visit were used to evaluate the occurrence of a transition from MCI to dementia according to DSM-V criteria.
  Chi square test for a 2x2 contingency table was used to compare patients who became demented at 1-year follow-up visit with those who did not, in the two treatment groups.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 21 | 22
Participants
  demented at 1-year follow-up | 3 | 5
  stable MCI | 17 | 17
  reverted to normal cognitive function | 1 | 0
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Test type: Superiority; p = .478, Chi-squared

9. Secondary Outcome: Cognitive Plasticity
Description: Improvement in long-term brain activity was measured by means of regional homogeneity (ReHo) of resting state functional MRI (rsfMRI) data. Statistical analysis of rsfMRI data was carried out by feeding Z-transformed ReHo data into voxel-wise inter-subject statistics using permutation-based nonparametric inference within the general linear model framework. P-values were calculated employing permutation-based statistics and corrected for multiple comparisons using the 3D parameter settings with threshold-free cluster enhancement, and a p-value <0.05 was considered statistically significant. Z-transformed ReHo differences (12 months-baseline) were computed separately for treated and non-treated patients, and a voxel-wise between-group comparison was used to evaluate the treatment effect . A positive mean of the Z-transformed ReHo differences represents an increase in activation over time (better outcome), and a negative mean represents a decrease in activation over time (worse outcome).
Time Frame: Baseline, 12 months
Population: RsfMRI data were available in in 22 patients (12 treated and 10 non-treated) after the exclusion of patients for technical reasons or head movement greater than 2 mm, and patients with incidental non-lacunar infarcts in the cerebral cortex, cerebellum, or brainstem to avoid a possible confounding effect on rsfMRI analysis.
Measure: Median (Inter-Quartile Range); unit: standard Z-values
Arm/Group | APT-II Group | Standard Care Group
Number analyzed (Participants) | 12 | 10
standard Z-values
  Z-transformed ReHo difference in vermis VIIIb | 0.78 [0.36 to 1.15] | -0.66 [-0.97 to -0.34]
  Z-transformed ReHo difference in right VIIb lobule | 1.02 [0.003 to 1.68] | -0.86 [-1.99 to -0.33]
  Z-transformed ReHo difference in left VIIb lobule | 1.31 [0.22 to 1.66] | -1.27 [-1.92 to -0.48]
Statistical Analysis 1: Comparison: APT-II Group vs Standard Care Group; Z-transformed ReHo difference in vermis VIIIb; Test type: Superiority; p = 0.029, General linear model voxel-wise — Corrected for multiple comparisons using the "3D" parameter settings with threshold-free cluster enhancement. A priori threshold for statistical significance 0.05
Statistical Analysis 2: Comparison: APT-II Group vs Standard Care Group; Z-transformed ReHo difference in right VIIb lobule; Test type: Superiority; p = 0.04, General linear model voxel-wise — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: APT-II Group vs Standard Care Group; Z-transformed ReHo difference in left VIIb lobule; Test type: Superiority; p = 0.039, General linear model voxel-wise — [p-value comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | APT-II Group | Standard Care Group
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APT-II Group (N=23) | Standard Care Group (N=23)
Cerebral haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes